CLINICAL TRIAL: NCT05738070
Title: Susceptibility Weighted Imaging for Detection of Thrombus in Acute Ischemic Stroke: a Cross-sectional Study.
Brief Title: Susceptibility Weighted Imaging for Detection of Thrombus in Acute Ischemic Stroke.
Status: Completed | Type: Observational
Sponsor: Upendra Devokta Memorial National Institute of Neurology and Allied Scicences (Other)
Responsible Party: Principal Investigator, Sushanta Paudel, Dr Sushanta Paudel, Upendra Devokta Memorial National Institute of Neurology and Allied Scicences
Other Study IDs: 113/2021
Record Dates: First submitted 2023-01-19; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Susceptibility vessel sign (SVS), MR angiography (MRA), thrombus length (TL)
MeSH Terms: conditions — Ischemic Stroke | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke: All the patients with stroke admitted to the hospital from July 2021 to July 2022 were included in this study. Patients with the following criteria were included in the study: (1) anterior circulation stroke established by diffusion-weighted imaging (DWI), (2) MRI performed within 72 hours of stroke onset, (3) Patient with occlusion of the vessel on MRA (Magnetic Resonance Angiography). (4) MRI performed before or during intravenous thrombolysis (IVT) or mechanical thrombectomy (MT). Infarcts with hemor¬rhagic transformation cases were not included in the study due to suboptimal SVS quantification
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — MRI was done in 1.5T unit (Siemens, Magnetom, Essenza). Different parameters for SWI as follows at 1.5T: echo time (TE) = 40 ms, repetition time (TR) = 29 ms, slice thickness = 0.7 mm, flip angle = 25°, field of view (FOV) = 184 × 200, intersection gap = 0 mm, and matrix size = 322 × 225. MRA parameters were as follows: TR = 29 ms, TE = 7.15 ms, FOV = 168 × 200 mm, slice thickness = 0.7 mm, flip angle = 25°, with acquisition time of 3 minutes.

SUMMARY:
It is a retrospective cross-sectional study, where consecutive stroke patients with vessel occlusion on magnetic resonance angiography (MRA) will be included for the study for one year. The relation of Susceptibility vascular sign (SVS) on Susceptibility Weighted Imaging (SWI) with risk factors and territory involved and length of thrombus will correlated with the National Institutes of Health stroke scale (NIHSS).Among total number of patients included in this study the demographics of the patients will be calculated. Risk factors for stroke of the patients included in this study will tabulated. The site of occlusion will be tabulated. The mean NIHSS scale will be calculated. Presence of SVS in patients with MR angiography positive vessel occlusion will be calculate in percentage. Subgroup analysis of presence of SVS on SWI will be done. The mean length of the thrombus will be calculated in these patients with positive SVS.

Correlation between SVS on SWI with the risk factor of the patient by using the chi-square test will be calculated. A Chi-square test will be done to find out the correlation between the SVS with territorial occlusion. The correlation between the NIHSS score and length of thrombus will be calculated using the Pearson test.

SWI can be useful in identifying the location of the thrombus, and NIHSS can determine the thrombus length in acute stroke. A higher incidence of SVS can be associated with risk factors and it also depends upon the site of occlusion of the vessel.

DETAILED DESCRIPTION:
Methodology:

This study will conducted at a tertiary level hospital with prior ethical approval from the institutional review committee and consent from the patient will taken with the consent form. It was a retrospective cross-sectional study design.

Patient selection: All the patients with stroke admitted to the hospital from July 2021 to July 2022 will included in this study. Patients with the following criteria will be included in the study: (1) anterior circulation stroke established by diffusion-weighted imaging (DWI), (2) MRI performed within 72 hours of stroke onset, (3) Patient with occlusion of the vessel on MRA (Magnetic Resonance Angiography). (4) MRI performed before or during intravenous thrombolysis (IVT) or mechanical thrombectomy (MT). Infarcts with hemor¬rhagic transformation cases were not included in the study due to suboptimal SVS quantification.

MRI Protocol: MRI will done in 1.5T unit (Siemens, Magnetom, Essenza). Different parameters for SWI as follows at 1.5T: echo time (TE) = 40 ms, repetition time (TR) = 29 ms, slice thickness = 0.7 mm, flip angle = 25°, field of view (FOV) = 184 × 200, intersection gap = 0 mm, and matrix size = 322 × 225. MRA parameters are as follows: TR = 29 ms, TE = 7.15 ms, FOV = 168 × 200 mm, slice thickness = 0.7 mm, flip angle = 25°, with acquisition time of 3 minutes.

Imaging analysis: Two blinded radiologists who are blinded to the clinical characteristics and other MRI images reviewed the SWI images independently. The criteria for detection of SVS as a hypointense signal within the artery on SWI is more than the size of the diameter of the homologous contralateral artery . The length of SVS within M1 MCA will be determined by the largest length of SVS at the particular slice. Signal loss within the vessel will termed vessel occlusion on MRA . A vascular neurointerventionists who will be blinded to the clinical characteristics and other MRI images will review the MRA for detection of vessel occlusion.

Statistics: The data will be analyzed in Statistical Package for Social Sciences (SPSS) software (ver. 21; IBM, Armonk, New York). The statistical value are significant when as p-value was <0.05. A Chi-square test will be done to find out the correlation between SVS on SWI with patient risk factors and SVS on SWI with territory involved. The correlation will be calculated between the size of the thrombus and the NIHSS score.

ELIGIBILITY:
Inclusion Criteria:

* Anterior circulation stroke established by diffusion-weighted imaging (DWI),
* MRI performed within 72 hours of stroke onset,
* Patient with occlusion of the vessel on MRA (Magnetic Resonance Angiography).
* MRI performed before or during intravenous thrombolysis (IVT) or mechanical thrombectomy (MT).

Exclusion Criteria:

• Infarcts with hemorrhagic transformation cases were not included in the study due to suboptimal SVS quantification.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with stroke admitted to the hospital from July 2021 to July 2022 were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Patients Demographics and risk factor | one year
  Among total number of patients included in this study patients will be assessed as name , age ,sex, risk factor. Risk factors for stroke of the patients included in this study will tabulated such as smoking, heart disease, alcohol etc .
Site of occlusion | one year
  The site of occlusion on Magnetic resonance angiography will be tabulated such as Middle cerebral artery, Anterior cerebral artery etc
Presence of SVS on SWI | one year
  Presence of Susceptible vascular sign (SVS) on susceptibility weighted imaging (SWI) in patients with MR angiography positive vessel occlusion will be calculate in percentage
Sub group analysis for positive susceptible vascular sign | one year
  Subgroup analysis of presence of SVS on SWI will be done as per site of occlusion , risk factor, age ,sex and mean thrombus length
Association of Positive SVS on SWI with Different factors | one year
  Chi-square test will be done to find out the correlation between the SVS with territorial occlusion and presence of SVS on SWI with the risk factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Sushanta Paudel, Bharatpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halefoglu AM, Yousem DM. Susceptibility weighted imaging: Clinical applications and future directions. World J Radiol. 2018 Apr 28;10(4):30-45. doi: 10.4329/wjr.v10.i4.30. PMID 29849962